CLINICAL TRIAL: NCT05860504
Title: Aetiology and Clinical Importance of Acute Cardiac Dysfunction in Critical Illness
Brief Title: Acute Cardiac Dysfunction in Critical Illnes
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jonatan Oras, Associate professor/Senior consultant, Sahlgrenska University Hospital
Other Study IDs: SCCCS
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Multi Organ Failure; Left Ventricular Dysfunction; Right Ventricular Dysfunction; Tako Tsubo Cardiomyopathy; Myocardial Infarction; Cardiomyopathy, Stress
MeSH Terms: conditions — Multiple Organ Failure; Ventricular Dysfunction, Left; Ventricular Dysfunction, Right; Takotsubo Cardiomyopathy; Myocardial Infarction | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal left ventricular systolic function: Patients with normal echocardiographic systolic function, defined as having left ventricular ejection fraction ≥ 50% and no regional hypokinesia
  Interventions: Diagnostic Test: Echocardiography
- Left ventricular dysfunction: Patients with echocardiographic left ventricular systolic dysfunction, defines as having left ventricular ejection fraction < 50% or left ventricular regional hypokinesia in at least two adjacent segments
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Cardiac magnetic resonance imaging; Diagnostic Test: Coronary CT

INTERVENTIONS:
Diagnostic Test: Echocardiography — All patients in the study will be examined with echocardiography
Diagnostic Test: Cardiac magnetic resonance imaging — Sub-group of patients with left ventricular systolic dysfunction will be examined with cMRI
  Other Names: cMRI
  Groups: Left ventricular dysfunction
Diagnostic Test: Coronary CT — Sub-group of patients with left ventricular systolic dysfunction will be examined with CCT
  Other Names: CCT
  Groups: Left ventricular dysfunction

SUMMARY:
The overall aim of the study is to establish the clinical importance of cardiac dysfunction, by estimating its incidence and impact on short- and long-term outcomes, in a mixed population of critically ill patients with multi-organ failure. Pathogenesis of cardiac dysfunction in critical illness and key molecules linked to this will be explored.

DETAILED DESCRIPTION:
During critical illness, the heart is exposed to extreme external stressors, which may contribute to heart failure. There is a lack of knowledge of what happens to the heart over the course of critical illness. The few studies available suggest that LV dysfunction is common in critical illness, with a prevalence of 10-30%. Notably, LV regional hypokinesia is a frequent pattern of LV dysfunction among these patients and is associated with a higher risk of death.

LV regional hypokinesia during critical illness may have several possible aetiologies, including ischemic, inflammatory or other/mixed processes. Of these, acute coronary artery obstruction is probably most important. Patients with sepsis, for example, and acute ST elevation myocardial infarction have twice the risk of death. Type II myocardial infarction can also lead to LV dysfunction due to insufficient coronary artery flow e.g., from tachycardia, hypotension and hypoxia, resulting in myocardial ischemia. In the absence of CAD, LV regional hypokinesia could also result from myocardial inflammation secondary to systemic inflammatory response, direct toxic effects of cytokines or pathogenic infiltration. Another possible aetiology is Takotsubo syndrome, an acute cardiac condition characterised by reversible regional hypokinesia, usually in the apical portion of the LV. The current paradigm suggests that Takotsubo syndrome is triggered by the overstimulation of the myocardium by catecholamines and is closely correlated to events involving severe emotional or physical stress. Cardiac dysfunction in critical illness is likely a phenotype of Takotsubo syndrome since patients in the ICU undergo extreme stress and are exposed to both endogenously-released and exogenously-administered catecholamines.

In critical illness, accurate diagnosis of LV dysfunction is challenging due to the similar clinical presentation of potential aetiologies. However, diagnosing the underlying aetiology of LV dysfunction is essential to provide appropriate treatment and optimise outcomes. CAD can be diagnosed with coronary angiography and cardiac computed tomography (CCT). In the absence of CAD, cMRI is useful. cMRI can differentiate between myocardial ischemia, and inflammation, as well as between an acute or past event.

In this study, patients are examined with echocardiography to identify those with cardiac dysfunction. In a sub-set of patients with LV dysfunction, patients will be examined with coronary CT (if no angiography performed) and cardiac MRI. Blood samples are collected for storage in biobank.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged > 18 years
2. Admitted to a participating ICU within 24 hours
3. Significant organ dysfunction involving at least two organ systems. This is defined as fulfilling both of the following:

   * At least 4 points on the SOFA scale (Sequential Organ Failure Assessment scale)
   * Having at least 1 point on the SOFA scale from at least two organ systems
4. Given informed consent from patient or permission to participate from next of kin

Exclusion Criteria:

1. Echocardiographic examination not possible (e.g., pneumothorax, draping etc) or very low echocardiographic examination quality
2. Not being examined with echocardiography within 24 hours from inclusion
3. Retracted consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant multi-organ dysfunction being admitted to a participaing ICU within 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 592 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
90-days mortality | 90 days
  Death

SECONDARY OUTCOMES:
Alive outside ICU | 90 days
  Days alive while not in the ICU
Alive without mechanical ventilation | 90 days
  Days alive and without mechanical ventilation
Alive without CRRT | 90 days
  Days alive without CRRT

CONTACTS AND LOCATIONS:
Locations (1):
- Sahgrensak University Hospital, Västra Frölunda, Please Select, Sweden